CLINICAL TRIAL: NCT04094779
Title: Effect of "breath of Fresh Air" Flash Activity on Dementia Agitation : Pilot Study
Acronym: DEMACTIFLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0348
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Dementia
Keywords: Agitation; Flash activity; Breath of fresh air
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual relational care (Active Comparator): Isolate the patient from the group of other patients in order to propose to him a a relationship dual with the caregiver to the aim to calm the agitation
  Interventions: Other: Usual relation care
- Flash activity "breath of fresh air" (Experimental): Isolate the patient from the group of other patients in order to propose to him in a relationship dual with the caregiver a physical activity outside the service that promotes relaxation by focusing his attention to the environment during 15 minutes
  Interventions: Other: Usual relation care; Other: Flash activity "breath of fresh air"

INTERVENTIONS:
Other: Usual relation care — When a patient begins to agitate, he will be isolated from the group to establish a dual relationship where the caregiver will try through his relational approach to calm the agitation.
Other: Flash activity "breath of fresh air" — When a patient begins to agitate , he will be isolated from the group and the patient leave from the unit to walk outside with the caregiver.
  Arms: Flash activity "breath of fresh air"

SUMMARY:
Non-drug therapies (NDT) constitute a strong axis of the person with dementia behaviour management. Among these NDT, the flash activities constitute a mode of intervention to prevent and control the expression of the most disruptive behavior. These are short-term activities with the objective of decreasing the behavioural disorders intensity in less than 15 minutes.

The aim of this pilot study is to test the effect of a flash activity "breath of fresh air" compared to the usual relational care on the short-term decrease (15 min.) of the agitation in hospitalized dementia patients.

DETAILED DESCRIPTION:
The "breath of fresh air" flash strategy is to offer the patient the possibility to go out of the medical unity and walking outdoor.

When the caregiver identify a level of agitation greater or equal to two on the gravity score and greater or equal to two on the impact score with the NPI test (The Neuropsychiatric Inventory Test), the caregiver let the patient wandering in the outside lanes of the hospital and encourage him to us his senses. For example, the sight could be stimulated by looking at a bird.

This variation of sensory stimulations enable a temporo-sensory break on the crisis, allowing the patient to turn his attention from the crisis context to another stimulation.

ELIGIBILITY:
Inclusion Criteria:

* New patients admitted in the unit to the management of the Psychological and Behavioural Symptoms of Dementia
* Dementia regardless of etiology and severity
* Score greater than 2 than NPI established on entry into service
* Free, informed and written consent signed by the person trust and/or family member and/or legal representative
* Health insurance membership

Exclusion Criteria:

* Absence of agitation
* Juveniles
* Pregnant women
* Patient who has previously participated in the study
* Persons under protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the NeuroPsychiatric Inventory Reduced (NPI-reduced) score | 15 minutes
  Evolution of the score NPI-reduced agitation 15 minutes after installation of the strategy compared to the score assessed in the crisis. NPI reduced is about Gravity of the crisis from1 to 3 (1 better / 3 worse) and Impact of the crisis from 0 to 5 (0 better / 5 worse)

SECONDARY OUTCOMES:
Comparison of the NPI-reduced score | 1 hours
  Evolution of the score NPI-reduced agitation 1 hours after installation of the strategy compared to the score assessed in the crisis. NPI reduced is about Gravity of the crisis from1 to 3 (1 better / 3 worse) and Impact of the crisis from 0 to 5 (0 better / 5 worse)
The Cohen-Mansfield Agitation Inventory (CMAI) score | 7 days
  Evaluation of the CMAI score to know the agitation level of the patient on the last 7 days with items about physical agitation and aggressivity, verbal agitation and aggressivity . From 0 to 203 (0 better / 203 worse)
The Cohen-Mansfield Agitation Inventory (CMAI) score | 18 days
  Evaluation of the CMAI score to know the agitation level of the patient on the last 18 days with items about physical agitation and aggressivity, verbal agitation and aggressivity . From 0 to 203 (0 better / 203 worse)
The NPI-CT (NeuroPsychiatric Inventory Care Team version) score | 21 days
  Evaluation oh the NPI-CT score to see the evolution of the overall intensity of behavioural disorders relative to the admission of patients. From 0 to 120 (0 better/ 120 worse)
Number of therapeutic strategies used | 18 days
  Number of therapeutic strategies (anxiolytics, hypnotic, neuroleptic or physical restraint) received at the outcome of an episode of agitation for which the "Breath of fresh air" in the experimental arm or the helping relationship in the arm control would have been insufficient

CONTACTS AND LOCATIONS:
Overall Officials: Aneta BARTUSIAK, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital Garonne, Toulouse, France

IPD SHARING:
Plan to Share IPD: No